CLINICAL TRIAL: NCT04062942
Title: The Six-Minute Walking Test (6WT) and Timed-Up-and-Go (TUG) Test as Measures of Objective Functional Impairment in Patients Undergoing Interlaminar or Transforaminal Epidural Steroid Injection for Lumbar Degenerative Disc Disease (DDD)
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: PD Dr. med. Martin Stienen, Klinik für Neurochirurgie, Universitätsspital Zürich (Unknown); PD Dr. med. David Bellut, Klinik für Neurochirurgie, Universitätsspital Zürich (Unknown); PD Dr. med. Oliver Gautschi, Neuro- und Wirbelsäulen Zentrum Zentralschweiz, Luzern (Unknown)
Responsible Party: Principal Investigator, Nicolai Maldaner, Principal Investigator, Cantonal Hospital of St. Gallen
Other Study IDs: OFI INJ - 1.0
Record Dates: First submitted 2019-08-17; First posted 2019-08-20 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Lumbar Disc Disease; Lumbar Spine Degeneration; Lumbar Spinal Stenosis
MeSH Terms: conditions — Intervertebral disc disease; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DDD patients: All patients presenting to the neurosurgical department of the Kantonsspital St. Gallen (KSSG) or the Univesity Hospital Zürich (USZ) with DDD fulfilling the inclusion criteria and scheduled for ESI or TFESI will be considered for this study.

SUMMARY:
The primary objective is to determine the validity of the Six-Minute-Walking Test (6WT) and Timed-Up and Go (TUG) test to measure objective functional impairment (OFI) in patients undergoing either interlaminar epidural steroid injection (ESI) or transforaminal epidural steroid injections (TFESI) for lumbar degenerative disc disease (DDD)

DETAILED DESCRIPTION:
The purposes of the project are to assess the ability of the Six-Minute-Walking Test (6WT) and Timed-Up and Go (TUG) test to measure and classify the disease burden, and to determine their relation to already established subjective patient reported outcome measures (PROMs)in patients treated with either interlaminar epidural steroid injection (ESI) or transforaminal epidural steroid injections (TFESI) for lumbar degenerative disc disease (DDD). No research has so far determined its validity to determine OFI in a cohort of patients managed conservatively. We want to use an existing smartphone-applications for the 6WT and TUG test. Applying self-measurement of the 6WT within the context of a two center observational study will determine OFI in patients before and after (TF)ESI. The results of this study add to the understanding of achievable objective outcomes after steroid injection applied to patients with DDD.

ELIGIBILITY:
Inclusion Criteria:

* Patient with symptomatic lumbar Degenerate Disc Disease (DDD), scheduled for either either interlaminar epidural steroid injection (ESI) or transforaminal epidural steroid injections (TFESI)
* Male and Female subjects ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Inability to walk (extreme pain or severe neurological deficits)
* Severe Chronic Obstructive Lung Disease (COPD) corresponding to ≥ Gold III
* Severe heart failure corresponding to ≥ New York Heart Association (NYHA) III
* Lung cancer and diffuse parenchymal lung disease
* Other medical reasons interfering with the patient's ability to walk and perform the 6WT/TUG (e.g., osteoarthritis disease of the lower extremities, Parkinson's disease, heart failure, hip or knee prosthesis etc.)
* Unavailability for follow up and/or inability to complete assessment (planning to move, no smartphone, etc.).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the neurosurgical department of the Kantonsspital St. Gallen (KSSG) or the Univesity Hospital Zürich (USZ) with DDD fulfilling the inclusion criteria and scheduled for ESI or TFESI will be considered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Raw Walking distance | 2-6 weeks
  The difference in 6WD (in m), as measured with the 6WT, between the baseline (before injection) and 4-week (range 2-6 weeks) follow-up assessment (after injection).

SECONDARY OUTCOMES:
Raw Walking distance - day 1 | 1 day
  Difference in Six-minute-walking test (6WD, in m) between baseline and 1-day follow-up
Raw Walking distance - day 7 | 7 days
  Difference in 6WD (in m) between baseline and 7-day follow-up
TTFS and DTFS - day 1 | 1 day
  Difference in Time to first symptoms (TTFS, in sec) and Distance to First Symptoms (DTFS, in m), as measured by the 6WT, between the baseline and 1-day follow-up assessment
TTFS and DTFS - day 7 | 7 days
  Difference in TTFS and DTFS, as measured by the 6WT, between the baseline and 7-days follow-up assessment
TTFS and DTFS - 4 weeks | 4 weeks
  Difference in TTFS and DTFS, as measured by the 6WT, between the baseline and 4 weeks follow-up assessment
ODI | 4 weeks
  Difference in PROM, as measured by the Oswestry Disability Index (ODI score, range 0% (best) - 100% (worst)), between the baseline- and 4-week follow-up assessment
COMI | 4 weeks
  Difference in PROM, as measured by the Core Outcome Measure Index (COMI score, range 0 (best) - 10 (worst)), between the baseline- and 4-week follow-up assessment
SF -12 | 4 weeks
  Difference in in health-related quality of life (hrQoL), as measured by the SF-12 score (SF-12 score, range 0 (worst) - 1 (best)), between the baseline- and 4-week follow-up assessment
NRS Pain | up to 4 weeks
  Difference in pain intensity, as measured by the NRS pain scale (NRS pain score, range 0 (best) - 10 (worst)), between the baseline- and 1-day, 7-day and 4-week follow-up assess-ments
Correlation 6WD/ODI | 4 weeks
  Correlation of 6WD with the ODI score at baseline and 4-week follow up
Correlation 6WD/COMI | 4 weeks
  Correlation of 6WD with the COMI score at baseline and 4-week follow up
Correlation 6WD/SF-12 | 4 weeks
  Correlation of 6WD with the SF-12 score at baseline and 4-week follow up
Correlation 6WD/NRS Pain | up to 4 weeks
  Correlation of 6WD with the NRS pain score at baseline and 1-day, 7-days and 4-week follow up
Correlation 6WD/TUG | 4 weeks
  Correlation of 6WD with the TUG test at baseline and 4-week follow up
TUG T-Score | 4 weeks
  Difference in TUG T-score between the baseline (before injection) and 4-week follow-up assessment (after injection)
Correlations TUG/PROMS | 4 weeks
  Correlation of TUG T-score with the ODI/COMI/NRS Pain/SF-12 score at baseline and follow up

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Maldaner, MD, Principal Investigator — Kantonsspital St. Gallen / Department of Neurosurgery; Martin Stienen, MD, Principal Investigator — Universitätsspital Zürich / Department of Neurosurgery
Locations (2):
- Switzerland (2):
  - Kantonsspital St. Gallen / Department of Neurosurgery, Sankt Gallen
  - University Hospital Zürich / Department of Neurosurgery, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stienen MN, Ho AL, Staartjes VE, Maldaner N, Veeravagu A, Desai A, Gautschi OP, Bellut D, Regli L, Ratliff JK, Park J. Objective measures of functional impairment for degenerative diseases of the lumbar spine: a systematic review of the literature. Spine J. 2019 Jul;19(7):1276-1293. doi: 10.1016/j.spinee.2019.02.014. Epub 2019 Mar 2. PMID 30831316
- [Result] Stienen MN, Maldaner N, Joswig H, Corniola MV, Bellut D, Prommel P, Regli L, Weyerbrock A, Schaller K, Gautschi OP. Objective functional assessment using the "Timed Up and Go" test in patients with lumbar spinal stenosis. Neurosurg Focus. 2019 May 1;46(5):E4. doi: 10.3171/2019.2.FOCUS18618. PMID 31042663